CLINICAL TRIAL: NCT01223209
Title: A Phase I, Combination, Immunologic Study of LTX-315 as Adjunct to GV1001 in Patients Following Curative Surgery for Carcinoma
Brief Title: A Study, Combination, Immunologic Study of LTX-315 as Adjunct to GV1001 in Patients Following Curative Surgery for Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lytix Biopharma AS (Industry)
Collaborators: Kael-GemVax Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: C09-315-02
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Carcinoma
Keywords: Cancer; Carcinoma; Curative surgery; Curative surgery for carcinoma at least three months and not more than 5 years prior to treatment start
MeSH Terms: conditions — Carcinoma; Neoplasms | interventions — LTX-315; GV1001 peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LTX-315 (Experimental): The dose range of 0,25-2.0 mg/ML LTX-315 will be used. In combination with a fixed dose of GV-1001.
  Interventions: Drug: LTX-315

INTERVENTIONS:
Drug: LTX-315 — 0.25-2.0 mg/ML, maximum 5 injections during 36 days.
  Other Names: GV-1001

SUMMARY:
This study involves testing of the medicine LTX-315 combined with a cancer vaccine (GV1001). This will be tested in patients that have had surgery with curative intent for malignant tumour.

GV1001 is a peptide vaccine in development to treat cancer. An adjuvant, is required to start the immune response in the body to have effect of GV-1001.

LTX-315, also a peptide, in development for cancer treatment. In this study, the investigators wish to find out whether LTX-315 can make GV1001 more effective at stimulating the immune system.

DETAILED DESCRIPTION:
This clinical study has two main aims which are:

* To measure the immunological effects of LTX-315 in combination with GV1001
* Find out about the side effects of the combination of the two drugs This is an open label, single centre study assessing immunological effects and safety of LTX-315 given as an adjunct to GV1001. The LTX-315 dose will escalate while the GV1001 dose will be fixed.

LTX-315 and GV1001 will be given as intradermal injections on days 1, 8, 15, 22 and 36.

Investigational treatment: LTX-315 (0.10 mL) with escalating concentrations will be injected intradermally, followed, 1-2 hours later, by intradermal injection of 0.56 mg GV1001 (0.20 mL, 2.8 mg/mL) in the same site, in one arm.

DTH-test control: 0.10 mg GV1001 (0.10 mL) will be injected intradermally in the contralateral arm without LTX-315, as a DTH skin reactivity test control.

ELIGIBILITY:
Inclusion Criteria:

* Curative surgery for carcinoma performed at least three months prior to treatment start
* Age ≥18 years
* ECOG Performance status (PS): 0
* Life expectancy: at least 3 months
* Laboratory requirements:

  * White Blood Count (WBC) ≥ 3 x 109/L
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Haemoglobin ≥ 10.0 g/dL
  * Total bilirubin level ≤ 1.5 ULN
  * AST and ALT ≤ 2.5 x ULN
  * Creatinine ≥ 1.5 ULN
  * Albumin > 30 g/L
* No expectation of anti-cancer therapy or immunotherapy during the trial period, hormone therapy given as adjunctive or contraceptive therapy is permitted
* Must be willing to practice acceptable barrier methods of birth control to prevent pregnancy
* The patient is willing and able to comply with the protocol and agrees to return to the hospital for follow-up visits and examination
* The patient has been fully informed about the study and has signed the informed consent form

Exclusion Criteria:

* Has received an investigational drug within 4 weeks prior to study drug administration, or is scheduled to receive one during the treatment or the post-treatment period
* Has received immunotherapy or been vaccinated within 12 weeks prior to study drug administration or has not recovered from adverse events due to such agents
* Has received external radiotherapy or cytotoxic chemotherapy within the last 4 weeks prior to study drug administration, or has not recovered from adverse events (< Grade 1) due to agents administered more than 4 weeks earlier
* Has received imiquimod within 12 weeks prior to study drug administration or has not recovered from associated adverse events
* Is currently on any agent with a known effect on the immune system
* Has any other serious illness or medical condition such as but not limited to:

  * Any uncontrolled infection or infection requiring antibiotics
  * Uncontrolled cardiac failure Classification III or IV (New York Heart Association)
  * Uncontrolled systemic and gastro-intestinal inflammatory conditions
  * Bone marrow dysplasia
  * History of auto-immune disease
  * History of adverse reaction to vaccines
* Known history of positive tests for HIV/AIDS, hepatitis B or C
* Is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Immunological effects of LTX-315 in combination with GV1001 as measured by DTH skin test reaction and T-cell function in peripheral blood. | 5 injections, treatment period 36 days
  Patients will return to the site 24 to 48 hours after the LTX-315 and GV1001 injections for DTH assessment and in week 10 for an end of study assessment.

SECONDARY OUTCOMES:
To evaluate the safety profile of LTX-315 in combination with GV1001 study | 5 injections, treatment period 36 days
  Assessment of adverse events and abnormal laboratory values recorded during the

CONTACTS AND LOCATIONS:
Overall Officials: Tone Nordøy, MD, PhD, Principal Investigator — Tromsø University Hospital
Locations (1):
- University Hospital North-Norway, Tromsø, Norway